CLINICAL TRIAL: NCT01245010
Title: Randomized Controlled Trial of a Water Beverage Intervention Trial for Reducing Risk Factors of Metabolic Syndrome in Young Mexican Free Living Women
Brief Title: Water Beverage Intervention Trial for Reducing Risk Factors of Metabolic Syndrome in Young Mexican Free Living Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mexican National Institute of Public Health (Other Government)
Collaborators: University of North Carolina, Chapel Hill (Other); Danone Global Research & Innovation Center (Industry)
Responsible Party: Principal Investigator, Sonia Hernandez-Cordero, Head of the Deparment of Community Nutrition, Mexican National Institute of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 755; CINYS 812 (Other: INSP)
Record Dates: First submitted 2010-05-20; First posted 2010-11-22 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Water; Obesity; Clinical trial; Prevention
MeSH Terms: conditions — Metabolic Syndrome; Obesity | interventions — Water; Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Water (Experimental): Water and education provision
  Interventions: Other: Water
- Control (Active Comparator): Education only
  Interventions: Other: Education

INTERVENTIONS:
Other: Water — Water and education will be provided
  Other Names: Water and education
  Arms: Water
Other: Education — Education
  Other Names: Education only
  Arms: Control

SUMMARY:
Research Question: Does replacing Sugar Sweetened (SS) beverages with water consumption promote a decrease in triglycerides blood levels over 9 months in overweight women? The primary outcome variable is the triglycerides blood level. In addition, the investigators will consider as secondary outcome variables the following parameters of metabolic syndrome: weight, fasting insulin and glucose, HOMA, HDL-cholesterol, systolic and diastolic blood pressure, and waist circumference. The investigators will also consider as an outcome variable glycosylated (or glycated) hemoglobin (HbA1c).

Design: Two groups randomized controlled trial, with an intervention group (water and education provision) and control group (education provision only).

The investigators propose to recruit young adult women aged >18-<45 y who are overweight or obese (BMI >25 and <39), and consume at least 250 calories per day from caloric beverages (e.g., includes soft drinks, juices, sports drinks, sweetened tea or coffee, and alcoholic beverages) The intervention group (water and education provision) will be compared with a control condition (education provision only). The intervention has been proposed to be carried out for 9 months period with objective measurements of body weight and fat, total cholesterol, LDL-C, HDL-C, fasting blood glucose, HbA1C, hydration status, blood pressure, and 24 hrs dietary recalls at baseline, 3,6 and 9 months

DETAILED DESCRIPTION:
Study subjects

The investigators propose to recruit young adult women aged 18-45 y who are overweight or obese (BMI >25 and <39), with fasting triglyceride level > 150 mg/dl, and consume at least 250 calories per day from caloric beverages (e.g., includes soft drinks, juices, sports drinks, sweetened tea or coffee, and alcoholic beverages). It is important to note that this is the average intake from caloric beverages for Mexican adolescent and adult women and represents the average Mexican adolescent and young woman behavior

Recruitment Participants will be recruited at a private weight-reduction clinic in Cuernavaca, Morelos (study site). Women will be invited to participate through local advertisements. Potential participants will be screened in order to evaluate if they fulfill the selection criteria of caloric beverages, BMI and triglyceride levels. Subsequently, in order to identify women with a high sweetened-beverage consumption women selected during the fist screening will be followed during a one-month period (referred to as the screening stage from now on), prior to recruitment into the intervention.

Screening stage This stage will consist in one month period of follow-up of women who have fulfilled the BMI, age, triglyceride and other selection criteria. During this period, three simplified 24-hr beverage-oriented dietary recalls (2 during week days and one weekend) will be collected approximately 7-10 days apart from each other. These 24 hr-recalls will exclusively seek to evaluate high caloric intake coming from sweetened caloric beverages. Specifically, the investigators will evaluate the consumption of all commercial and homemade caloric sweetened beverages (including juices, "aguas frescas", coffee and tea with added sugar). The investigators will also measure triglyceride levels in a blood drop collected through finger prick, at the study site. The specimen collection process will be quick, and with minimal discomfort for the participants. The investigators will use special lancet and a couple of drops of blood will be taken from a nick of a finger and deposited onto special analytic strip. Finally, a pregnancy test will be performed at the first visit for confirmation purposes.

Upon conclusion of the screening stage eligible participants will be randomly assigned to either the intervention or control group.

Given that the intervention will require participant's time involvement, throughout the intervention period all participants will receive a $15 compensation plus snacks at each follow-up visit. This sum was established based on the estimated cost of a time taken for work to attend visits and the cost of transportation to and from the clinic.

The Intervention

The intervention group (water provision) will be compared with a control condition (control group). The intervention has been proposed to be carried out for 9 months period with objective measurements of body weight and fat, total cholesterol, LDL-C, HDL-C, fasting blood glucose, HbA1C, hydration status, blood pressure, and 24 hrs dietary recalls at baseline, 3,6 and 9 months. Body weight will be also assessed at other times during the study. Eligible subjects, identified during the screening stage, will be randomly assigned either to receive water or to the control group. Boyh groups will be identical in all, except for the water deliveries and promotion of reducing the intake of sweetened caloric beverage and their substitution by an increase in water promotion. In order to pursuing this, specific counseling targeting to rationale and strategies for replacing caloric beverages to promote weight loss will be provided to the intervention group. In order to ensure that participants are not aware to the study group which they belong to (intervention or control group), the investigators will provide both groups with the same counseling in nutrition topics, except regarding the water consumption information.

Intervention description (Water group) and contacts: The goal for subjects assigned in the water group will be to reduce to a minimum or null the intake of caloric beverages, including carbonated (fizzy) and non-carbonated (still) beverages, coffee and tea with sugar, milk or cream added, juice drinks, soy beverages, and sugar sweetened "aguas frescas", , energy drinks, and smoothies. Participants will be instructed to drink water, replacing the caloric beverages mentioned above. Subjects assigned to this group will receive biweekly home deliveries of water during the 9 month of the intervention period.

In order to answer the research questions outlined above, adherence to the beverage reduction recommendations must be strongly promoted. To support the modification of beverage intake in the intervention group, participants will take part on monthly face to face treatment meetings will be held with trained dietician and or weight loss interventionists. These meetings will be held at convenient times and will be conducted on an individual basis as well as for groups of 8 to 10 participants . Participants will be weighed at each monthly meeting and weekly beverage consumption data will be collected. The individual and group meetings will cover rationale and strategies for replacing caloric beverages to promote weight loss. During the meetings challenges associated with the proposed behavior change and potential solutions will be discussed, and behavioral modification strategies to promote compliance will also be addressed. In addition, the weight loss interventionists and/or trained dieticians will call participants in a biweekly basis in order to maintain enthusiasm, ask for water supply status, and help solving challenges faced during the week.

Water/Beverage Provision:

To insure water availability, bottled water will be home delivered during the intervention period and/or available for pick-up at the monthly follow-up visits. Based on the work of Ebbeling et al.( ), the investigators plan to provide between 2 to 3 liters of water per person per day with 2 additional servings per day being provided to account for possible consumption of other family members, though this will be discouraged. Another option the investigators have identified in order to address the issue of consumption of the water provided by other family members is to provide an additional water dispenser for the household and additional large bottle of water for participants. The investigators will insure that participants receive the adequate serving sizes to fit their needs, for instance adequate bottle size to take water to workplace or other places. The qualitative component of the study will allow us to ascertain the size and number of water bottles to be provide to each participant.

In addition, the investigators will meet with the Bonafont, Mexico, marketing team to discuss how consumers use water and bottle size issues. This will be invaluable not only in the selection of beverage sizes but also in the design of the water consumption nutrition promotion programs.

Control group and contacts: Like the water group, the subjects in the control group will receive general nutrition advice not related to weight or food intake. They will not be granted specific information on reducing caloric beverage intake information related to beverage consumption and health. Participants in this group will be contacted following the same contact schedule and frequency as intervention group participants.

ELIGIBILITY:
Inclusion Criteria:

* Young adult women aged >18-<45 y
* BMI >25 and <39
* Consume at least 250 calories per day from caloric beverage
* Women planning to live in the study area over the next year
* Willingness to participate in the required evaluations
* Women have given their consent to participate

Exclusion Criteria:

* Report losing >5% of current body weight in the previous 6 months. Individuals who have recently lost significant body weight may be at high risk for weight regain, which could result in this study examining prevention of weight regain rather than weight loss.
* If they report to be on a diet to reduce weight at the time of recruitment
* Report pregnancy during the previous 6 months or if they are lactating at the time of recruitment or they are planning to become pregnant in the following 12 months.
* Report current treatment for any medical condition that could impact metabolic function (e.g.., diabetes mellitus, cancer, Etc.).
* History of myocardial infarction or heart surgery such as bypass or angioplasty. These individuals will be excluded because this may require additional medical monitoring and adjustments to the exercise prescription.
* Report taking any type of medication that could affect metabolism, energy intake or change body weight (e.g., hypothyroidism).
* Report hospitalization for psychiatric problems prior year to the enrollment period.
* If they are on a regime to increase muscle mass or taking anabolics
* Excessive consumption of alcoholic beverages, defined as 21 or more drinks per week

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2009-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Triglycerides blood level | baseline
Triglycerides blood levels | 3 months
Triglycerides blood Levels | 6 months
Triglycerides blood levels | 9 months

SECONDARY OUTCOMES:
Body weight | Baseline
Fasting insulin | Baseline
Fasting glucose | Baseline
Homeostasis Model Assessment (HOMA) | Baseline
HDL-cholesterol | Baseline
Systolic and diastolic blood pressure | Baseline
Waist circumference | Baseline
Glycosylated (or glycated) hemoglobin (HbA1c) | Baseline
Boby Weight | 3 months
Body weight | 6 months
Body weight | 9 months
Fasting insulin | 3 months
Fasting insulin | 6 months
Fasting insulin | 9 months
Fasting glucose | 3 months
Fasting glucose | 6 months
Fasting glucose | 9 months
Homeostasis Model Assessment (HOMA) | 3 months
Homeostasis Model Assessment (HOMA) | 6 months
Homeostasis Model Assessment (HOMA) | 9 months
HDL-cholesterol | 3 months
HDL-cholesterol | 6 months
HDL-cholesterol | 9 months
Systolic and diastolic blood pressure | 3 months
Systolic and diastolic blood pressure | 6 months
Systolic and diastolic blood pressure | 9 months
Waist circumference | 3 months
Waist circumference | 6 months
Waist circumference | 9 months
Glycosylated (or glycated) hemoglobin (HbA1c) | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Public Health, Cuernavaca, Morelos, Mexico

REFERENCES:
- [Derived] Rodriguez-Ramirez S, Gonzalez de Cosio T, Mendez MA, Tucker KL, Mendez-Ramirez I, Hernandez-Cordero S, Popkin BM. A Water and Education Provision Intervention Modifies the Diet in Overweight Mexican Women in a Randomized Controlled Trial. J Nutr. 2015 Aug;145(8):1892-9. doi: 10.3945/jn.115.212852. Epub 2015 Jul 1. PMID 26136584
- [Derived] Hernandez-Cordero S, Barquera S, Rodriguez-Ramirez S, Villanueva-Borbolla MA, Gonzalez de Cossio T, Dommarco JR, Popkin B. Substituting water for sugar-sweetened beverages reduces circulating triglycerides and the prevalence of metabolic syndrome in obese but not in overweight Mexican women in a randomized controlled trial. J Nutr. 2014 Nov;144(11):1742-52. doi: 10.3945/jn.114.193490. Epub 2014 Sep 3. PMID 25332472